CLINICAL TRIAL: NCT04726514
Title: SleepFlexTM Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berendo Scientific, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0100
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SleepFlex Treatment (Experimental)
  Interventions: Device: SleepFlex

INTERVENTIONS:
Device: SleepFlex — SleepFlex Program

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the SleepFlex program for treatment of mild to moderate OSA

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Mild to moderate OSA, defined as AHI >10 - 30 events/hour, documented by polysomnogram or home sleep apnea test within 180 days prior to study enrollment
* Central or mixed disordered breathing events (≤25% of total number of events)
* Unable to tolerate or decline positive airway pressure therapy
* Body mass index ≤32 kg/m2
* Able to protrude tongue ≥20 mm beyond maxillary incisors
* Absence of markedly enlarged tonsils, defined as 3+ or 4+ according to the Brodsky classification
* No uncontrolled sleep disorder other than OSA such as narcolepsy, chronic insomnia, restless legs syndrome, or REM behavior disorder
* Absence of excessive daytime sleepiness, defined by Epworth Sleepiness Scale score >10
* No uncontrolled nasal obstruction
* Absence of moderate to severe mandibular insufficiency
* No previous surgery involving the oral cavity or pharynx other than tonsillectomy
* No previous radiation therapy to the head and neck
* No known neurologic, cardiac (other than hypertension controlled with a single medication), pulmonary, renal, hepatic, or psychiatric disorders
* No psychiatric diagnoses other than treated depression or mild anxiety
* Stable medication regimen for ≥1 month
* No acute illness or infection
* Ownership of personal smartphone with iOS or Android operating system
* No known hypersensitivity to any material of the SleepFlex devices

Exclusion Criteria:

* Unwilling or unable to provide informed written consent in English
* Pregnancy, breastfeeding, or plans to become pregnant
* Smoker (tobacco or recreational drugs) in the past month
* Alcohol consumption, averaged over the previous month, greater than 2 alcoholic beverages per day
* Significant vision or hearing problems
* Unwilling or incapable of returning for all follow-up visits and conduct sleep studies at home, including the evaluation procedures and filling out questionnaires
* Any other reason the investigator determines as being unfit for study participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tower Sleep Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical office
Period: Overall Study
Arm/Group | SleepFlex Treatment
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
apnea-hypopnea index [Mean (Standard Deviation); unit: events/hour] — The apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. Apneas are defined by >=80% reduction in airflow for >= 10 seconds in the presence of respiratory effort. Hypopneas are defined by >=50% reduction in airflow with oxygen desaturation of >=3% in the presence of respiratory effort. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe. It was measured on a pre-treatment home sleep apnea test performed after study enrollment.
  events/hour | 15.1 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From SleepFlex-related Serious Adverse Events
Description: Number of participants with absence of serious adverse events related to the SleepFlex system.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Change in the Apnea-hypopnea Index (AHI)
Description: Change in the apnea-hypopnea index (AHI) on post-treatment vs. pre-treatment home sleep apnea test. Apneas are defined by >=80% reduction in airflow for >= 10 seconds in the presence of respiratory effort. Hypopneas are defined by >=50% reduction in airflow with oxygen desaturation of >=3% in the presence of respiratory effort. The Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of recording time. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 7
events/hour | 2.9 (3.5)

3. Secondary Outcome: Number of Participants With Development of Side Effects: Mouth, Throat, or Neck Pain; Dysphagia
Description: Number of participants with development of the following potential side effects: mouth, throat, or neck pain; dysphagia. This was assessed repeatedly throughout the study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 10
Participants | 0

4. Other Pre Specified Outcome: Change in Supine AHI
Description: Change in the supine apnea-hypopnea index (AHI) on post-treatment vs. pre-treatment home sleep apnea test.The Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe. The supine position is defined by sleeping on one's back.
Time Frame: 12 weeks
Population: Participants who completed study
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 7
events/hour | 5.7 (6.1)

5. Other Pre Specified Outcome: Change in Non-supine AHI
Description: Change in the non-supine apnea-hypopnea index (AHI) on post-treatment vs. pre-treatment home sleep apnea test.The Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe. The non-supine position is defined by sleeping in body positions other than one's back. Body position information is collected by the home sleep apnea test, and position-specific information is calculated.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | SleepFlex Treatment
Number analyzed (Participants) | 7
events/hour | 0.5 (4.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SleepFlex Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04726514/Prot_SAP_001.pdf